CLINICAL TRIAL: NCT05717972
Title: Effects of Kombucha Intervention on Emotional Distress and Sleep Quality in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, I-Ching Hou, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YM111146EF
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Distress, Emotional; Sleep
MeSH Terms: interventions — Kombucha Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Experimental)
  Interventions: Other: Kombucha
- B Group (Other): Waiting list
  Interventions: Other: Kombucha

INTERVENTIONS:
Other: Kombucha — Kombucha is a fermented tea drink that originated in ancient Chinese civilization. It is made by combining tea, juice, and SCOBY (Symbiotic Culture of Bacteria and Yeast).
  During the fermentation process, the yeast in the SCOBY breaks down the sugar in the tea releasing friendly probiotic bacteria, giving kombucha its fizzy body and its sweet and tangy taste.

SUMMARY:
Effects of Kombucha Intervention on Emotional Distress and Sleep Quality in Breast Cancer Survivors.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III Breast Cancer
* No any cancer treatment in the following year
* Perceived emotional distress and poor sleep quality
* Agree to follow the protocol of this study

Exclusion Criteria:

* Stage IV Breast Cancer
* Pregnant women
* Abnormal liver, kidney, gastric, internal , immune, sleep disorder, metabolic, psychic functions and need to take the prescription medications or medical treatments regularly
* could not follow the protocol of this study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality Index | Change from Baseline Sleep Quality Index at Day 20
  The Pittsburgh Sleep Quality Index, PSQI. The range of score was 0-21. The higher score and the worse sleep quality.
Sleep Quality Index | Change from Baseline Sleep Quality Index at Day32
  The Pittsburgh Sleep Quality Index, PSQI. The range of score was 0-21. The higher score and the worse sleep quality.
Anxiety | Change from Baseline State-Trait Anxiety Inventory at Day20
  The State-Trait Anxiety Inventory, STAI. It includes two types of anxiety. The state anxiety is considered to be individual's temporary perception toward fear, nervousness, discomfort etc. and the trait anxiety be the individual's experience on a daily basis The range of each measurement score was 20-80. Higher scores indicate greater anxiety.
Anxiety | Change from Baseline State-Trait Anxiety Inventory at Day32
  The State-Trait Anxiety Inventory, STAI. It includes two types of anxiety. The state anxiety is considered to be individual's temporary perception toward fear, nervousness, discomfort etc. and the trait anxiety be the individual's experience on a daily basis The range of each measurement score was 20-80. Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 2
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 3
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 4
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 5
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 6
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 7
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 8
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 9
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 10
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 11
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 12
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 13
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 14
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 15
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 16
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 17
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 18
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 19
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 20
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 21
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 22
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 23
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 24
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 25
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Intestinal Transit Time | Change from Baseline Bristol Stool Form Scale at Day 26
  Bristol Stool Form Scale, BSFS. It is a useful guide to intestinal transit time by describing the shapes and types of stools(type 1 to 7).
  Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.

CONTACTS AND LOCATIONS:
Overall Officials: I-Ching Hou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided